CLINICAL TRIAL: NCT04973891
Title: Canagliflozin Administration in Non-diabetic Women With Polycystic Ovarian Syndrome
Brief Title: CANA/Met in Non-diabetic Women With PCOS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Bing He, Professor Bing He, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 777
Record Dates: First submitted 2021-07-09; First posted 2021-07-22 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Canagliflozin/metformin group (Experimental): Intervention with canagliflozin combined with metformin for three months
  Interventions: Drug: Canagliflozin combined with metformin
- Active Comparator: Metformin group (Active Comparator): Intervention with metformin for three months
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: Canagliflozin combined with metformin — Canagliflozin, a novel glucose-lowering medication, has been shown to have positive effects on reducing body weight, blood pressure and cardiovascular events.
  Metformin, a classical and common insulin sensitizer that can reduce both hyperinsulinemia and hyperandrogenemia, is widely used for patients with PCOS.
  Arms: Experimental: Canagliflozin/metformin group
Drug: metformin — Metformin, a classical and common insulin sensitizer that can reduce both hyperinsulinemia and hyperandrogenemia, is widely used for patients with PCOS.
  Arms: Active Comparator: Metformin group

SUMMARY:
Polycystic ovary syndrome (PCOS), which is associated with hyperinsulinaemia, hyperandrogenaemia, impaired glucose metabolism and aberrant adipokines production from the adipose tissue, is a heterogeneous reproductive and endocrine disorder.Currently, metformin, a classical and common insulin sensitizer that can reduce both hyperinsulinemia and hyperandrogenemia, is widely used for patients with PCOS. SGLT-2 inhibitor, a novel glucose-lowering medication, have been shown to have positive effects on reducing body weight, blood pressure and cardiovascular events in individuals with diabetes mellitus. However, evidences related to its management in non-diabetic PCOS women are limited. Hence, we want to give canangliflozin combined with metformin to women with PCOS to see its effect on insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18- 45 years old;
2. Diagnosed criteria meet the Rotterdam criteria (2003);
3. Insulin Resistance

Exclusion Criteria:

1. Women who are pregnant or have a pregnancy plan within six months;
2. Confirmed diagnosis of diabetes.
3. Congenital adrenocortical hyperplasia;
4. Hyperprolactinemia;
5. Hyperthyroidism or hypothyroidism;
6. Combined with liver or kidney diseases;
7. Abnormal liver function (≥ 3 times of the upper limit of normal range);
8. Abnormal renal function (GFR<60ml/min/1.73m2);
9. Adrenal or ovarian tumors secreting androgens;
10. Used metformin, glucagon-like peptide-1 receptor agonists, pioglitazone and contraceptives in the last 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Body mass index | Three months
  Changes in body mass index (BMI)

SECONDARY OUTCOMES:
Total testosterone | Three months
  Changes in total testosterone (TT)
Androstenedione | Three months
  Changes in androstenedione (AND)
Dehydroepiandrosterone sulfate | Three months
  Changes in dehydroepiandrosterone sulfate (DHEA-S)
Sex hormone-binding globulin | Three months
  Changes in sex hormone-binding globulin (SHBG)

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Zhang J, Xing C, Cheng X, He B. Canagliflozin combined with metformin versus metformin monotherapy for endocrine and metabolic profiles in overweight and obese women with polycystic ovary syndrome: A single-center, open-labeled prospective randomized controlled trial. Front Endocrinol (Lausanne). 2022 Sep 6;13:1003238. doi: 10.3389/fendo.2022.1003238. eCollection 2022. PMID 36147577